CLINICAL TRIAL: NCT01765517
Title: A 26-week, Randomized, Double-blind, Placebo-controlled Study to Explore the Effects of Probiotics on Endotoxin Levels in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Explore the Effects of Probiotics on Endotoxin Levels in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Warwick Medical School (Other); Winclove Bio Industries BV (Industry)
Responsible Party: Principal Investigator, Nasser Al-Daghri, Professor, King Saud University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11-MED2114-02; NPST_Alokail (Other Grant/Funding Number: NPST)
Record Dates: First submitted 2013-01-01; First posted 2013-01-10 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): Probitoics
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Administration of probiotics daily for 26 weeks and compared to placebo
  Other Names: Ecologic Metabolic
  Arms: Probiotics
Dietary Supplement: Placebo — Administration of placebo daily for 26 weeks and compared to probiotics group
  Arms: Placebo

SUMMARY:
Probiotics, which are believed to be health promoting live microorganisms, have been reported to influence circulating endotoxin levels. Ingestion of the live cultures may alter gut mircobiota in a beneficial manner to reduce inflammation; although their mechanism and influence to reduce inflammation in T2DM is not established for this disease state. Therefore, the aim of this study is to (1) characterize the beneficial effects of probiotics on circulating endotoxin levels and other biomarkers related to systemic low-grade inflammation in patients with T2DM; (2) Compare circulating endotoxin levels and inflammatory cytokine levels between patients treated with probiotics or placebo to examine the beneficial effects of probiotics on reducing the inflammatory status, through assessment of systemic markers (adipokines, endotoxin, cytokines); (3) to examine the effects of probiotics on gut microflora in order to understand the mechanism for such change in inflammatory status. To achieve this, 120 consenting adult Saudis, naïve or newly diagnosed T2DM patients without co-morbidities, will be enrolled in this clinical trial and randomized to receive twice-daily placebo or probiotics for 26 weeks in a double-blind manner. Glycemic inflammatory markers will be measured and fecal samples analysed, interventions will be done at baseline, 4, 8, 12 and 26 weeks. It is envisaged that probiotics will induce beneficial changes in gut mircobiota, reduce the systemic inflammatory state through altering systemic endotoxin levels and, as such, reduce the systemic inflammatory response observed in T2DM subjects. This will have a fundamental impact on how we should treat the inflammatory component of T2DM, particularly once the results are verified in a larger cohort of patients, as this could have very dramatic effects on how we treat patients with T2DM. Reducing the pathogenesis of T2DM by dampening the inflammatory response, which may also impact on insulin resistance status and health of the individual, will have clear benefits. This could have profound effects on preventative T2DM management, as well as current T2DM care without excessive cost for the wider Saudi health economy.

DETAILED DESCRIPTION:
Design

In this 26-week, single-center, double-blind, randomized, placebo-controlled study, 60 patients with T2DM will be treated with probiotics and 60 will be treated with placebo. Interventions will be done at weeks 0, 4, 8, 12 and 26 from all subjects. Patients allocated to the probiotics group will receive capsules containing four strains of freeze-dried bacteria, namely Lactobacillus acidophilus, Lactobacillus bulgaricus, Bifidobacterium bifidum, and Streptococcus thermophiles (Bio-plus®, Supherb, Israel), at a daily dose of 2 × 1010 CFU. Participants in the placebo group will receive capsules containing wheat-based non-fermentable fibers, as used in another clinical trial [Pereg et al, 2011].

Recruitment of Patients

Recruitment of patients to this study will be made possible by collaboration with primary care centers throughout Riyadh and the Biomarkers Research Program, College of Science, King Saud University.

Inclusion Criteria

* Stable and well controlled T2DM (HbA1c < 7.5% and no change in oral antidiabetic medications during the last 6 months)
* Age 20-75 years
* Provision of written informed consent

Exclusion Criteria

* Chronic gastrointestinal disease (except IBS)
* Systemic antibiotics within 6 weeks before inclusion
* Use of probiotics within 3 months before inclusion (Appendix A lists products currently marketed internationally and available to purchase in Saudi Arabia)
* Regular intake of insulin or insulin analogs, antibiotics or probiotics, antacids, H2-receptor blockers, proton pump inhibiters, loperamide, cholestryramine, ω3 supplements, fibrates, corticosteroids or sex steroids
* Daily alcohol consumption > 30 g
* Significant immunodeficiency
* Known cardiac valvular disease
* Breast-feeding or pregnant
* Non-Arab ethnicity
* Participation in another clinical trial within the last 6 months
* Legal incapability

Allocation to Treatment

After confirmation of eligibility and obtaining written informed consent, the patients will be given a unique subject number by the probiotics company, who also will perform the randomization (stratified for gender), The patients and clinicians at the primary care center will be blinded to the treatment received. The eligible patients will be allocated (1:1) to treatment for 26 weeks with either the probiotics supplement or placebo. Subjects will be instructed to

* Ingest 1 capsule before breakfast and 1 capsule before the evening meal, either directly or mixed in standard yoghurt.
* The capsules will be stored in the refrigerator after the jar has been opened.

Data Handling and Record Keeping

Case report form (CRF) will be used to record data for all participants, and will be completed by the research nurse, who will also enter the data into an electronic database.

Study schedule and location

After inclusion, all further treatments will be managed at the primary care center where the subject was recruited (see appendix C for scheduled visits). A research nurse and a research dietician will be responsible for all contact with patients. Doctors associated with the research team will be available if problems arise.

Acquisition of Clinical Data and Assessment of Compliance

* Medical history, including the presence of chronic diseases, regular medication, smoking and alcohol habits, will be recorded before inclusion.
* Nutritional habits will be assessed using a standardized 14-day recall questionnaire, which will be discussed with a dietician
* Changes in medication during the study period will be recorded
* Anthropometric measurements will be made using standardized methods. Height will be measured at the start of treatment. Weight (in light clothing without shoes or items in pockets), waist circumference (measured as a horizontal plane at the level of the umbilicus) and hip circumference (measured as a horizontal plane at the level of the trochanter major) will be measured at the start and end of the treatment.
* Liver ultrasonography will be performed either at screening or at the start of treatment to determine the presence or absence of a bright liver indicative of steatosis. Patients with fatty liver and liver transaminases > 1.5 × the upper limit of normal will be offered referral to a hepatologist.
* Compliance will be monitored at weeks 4, 8, 12 and 26. Patients will bring their previously received capsules to the primary care center to calculate the mean number of capsules ingested per day.

Acquisition of Routine Biochemical Data and Biological Samples

* Blood samples obtained will be analyzed at the Biomarkers Research Program to measure glucose, HbA1c, insulin, C-peptide, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, alanine aminotransferase and aspartate aminotransferase levels.
* Fasting blood samples will be collected at week 0, 8 and 26. Peripheral venous blood will be drawn into pyrogen-free tubes without any anticoagulant. The tubes will be immediately placed in ice, allowed to coagulate, and centrifuged (2500 ×g for 10 min at 4°C) within 2 hours of collection. Serum samples will be stored at -80°C until use. At least two 2-mL serum samples will be collected at each time-point.
* Stool samples will be taken by asking patients to store the sample in a plastic sealable bag in their freezer until transfer to the clinic. (samples taken at the same points as they are requested for blood samples. Once at the clinic, the samples will be divided, flash frozen, and stored at -80°C. Changes in gut microbiota will be profiled using signature-tagged sequencing (pyrosequencing) of amplified 16S rRNA genes followed by automated bioinformatics analysis. Targeted RT-PCR will also be used to examine bacterial species such as Enterobacteria and Bifdobacteria relative to the universal bacterial primer set. Pyrosequencing and RT-PCR will be performed in a sub-cohort (n=15) of patients considering the final systemic findings. Samples will be retained for subsequent studies.

Subject Withdrawal

Subjects may withdraw from the trial at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator for safety, behavioral or administrative reasons. The subjects will also be withdrawn from the study in case of:

* Treatment with systemic antibiotics for > 1 weeks during week 0-22
* Any use of systemic antibiotics during week 22-26

Patient Safety

Adverse Events

Adverse events (AEs) are undesirable signs or symptoms that occur during the study and may or may not be causally related to the treatment. All AEs considered possibly, probably or definitely related to the test product will be recorded on CRFs.

Serious Adverse Events

Serious adverse events (SAEs) are defined as events that are fatal, life-threatening, disabling, incapacitating or result in hospitalization or prolong hospital stay, or result in malformation. All SAEs will be recorded in the CRF, whether they are related to the test product or not. According to previous studies (9), probiotics are very safe, and any SAE that might be possibly, probably or definitely related to the test product will be regarded as unexpected. All unexpected SAEs will be reported immediately to the Medicines and Healthcare products Regulatory Agency (MHRA). Any SAE that might be related to the test will immediately lead to discontinuation of the test product.

Ethical and Regulatory Aspects

The study will be performed in accordance with the protocol and the ethical principles that have their origin in the Declaration of Helsinki as well as with the International Council for Harmonization Guidance on Good Clinical Practice. These documents state that the informed consent of subjects is an essential precondition for participation in the clinical study. The study will commence only after obtaining approval from the local ethical review board of the College of Medicine Research Center, King Saud University.

Plan for Data Analyses

As this trial is designed to assess the physiological effects rather than support clinical indications for treatment with probiotics in T2DM, we plan to perform per protocol analyses. Only subjects treated with at least 80% of the planned doses for at least 80% of the time will be considered as treated per protocol.

Raw data will be entered in a statistical software (Statistical Package for the Social Sciences), SPSS version 16.5 (Chicago, IL, USA). Preparation of data set will be done prior to analyses. Descriptive statistics will be done; frequencies will be presented in percentage (%). Continuous variables will be presented as mean ± standard deviation. Variables exhibiting non-Gaussian variables will be transformed prior to analyses. Repeated measures analysis of co-variance (ANCOVA) will be used to compare groups, which will represent a combination of analysis of variance (ANOVA) and linear regression. Confounding and fixed variables such as age and gender, as well as BMI will be taken if proper matching has not been achieved prior to repeated measures. Post-hoc Banjamini-Hohberg corrections will be done for multiple comparisons. For comparison of 2 groups, independent T-test will be done for continuous variables and Mann-Whitney for non-continuous variables. Analysis of adverse events (if any) will be done using Chi-Square test and Fisher's exact test following assumptions of randomness, independence and size. Significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Stable and well controlled T2DM (HbA1c < 7.5% and no change in oral antidiabetic medications during the last 6 months)
* Age 20-75 years
* Provision of written informed consent

Exclusion Criteria:

* Chronic gastrointestinal disease (except IBS)
* Systemic antibiotics within 6 weeks before inclusion
* Use of probiotics within 3 months before inclusion (Appendix A lists products currently marketed internationally and available to purchase in Saudi Arabia)
* Regular intake of insulin or insulin analogs, antibiotics or probiotics, antacids, H2-receptor blockers, proton pump inhibiters, loperamide, cholestryramine, ω3 supplements, fibrates, corticosteroids or sex steroids
* Daily alcohol consumption > 30 g
* Significant immunodeficiency
* Known cardiac valvular disease
* Breast-feeding or pregnant
* Non-Arab ethnicity
* Participation in another clinical trial within the last 6 months
* Legal incapability

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
effects of probiotics on endotoxin levels in patients with T2DM | 1 year
  Exploration of baseline characteristics and determination of associations between nutritional habits, gut flora and levels of endotoxin/inflammatory markers at baseline and subsequent follow ups

SECONDARY OUTCOMES:
effects of probiotics on gut microflora | 1 year
  Determine changes from baseline in the amount of probiotics, all anaerobic bacteria and short-chain fatty acids (e.g., propionate and butyrate) present in fecal samples.

OTHER OUTCOMES:
Effects of probiotics on insulin resistance | 1 year
  Determine changes from baseline in serum levels of glucose, HbA1C, insulin and C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Al-Daghri, PhD, Study Chair — King Saud University; Majed Alokail, PhD, Principal Investigator — King Saud University
Locations (1):
- Biomarkers Research Program, King Saud university, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Sabico S, Al-Mashharawi A, Al-Daghri NM, Wani K, Amer OE, Hussain DS, Ahmed Ansari MG, Masoud MS, Alokail MS, McTernan PG. Effects of a 6-month multi-strain probiotics supplementation in endotoxemic, inflammatory and cardiometabolic status of T2DM patients: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2019 Aug;38(4):1561-1569. doi: 10.1016/j.clnu.2018.08.009. Epub 2018 Aug 17. PMID 30170781
- [Derived] Sabico S, Al-Mashharawi A, Al-Daghri NM, Yakout S, Alnaami AM, Alokail MS, McTernan PG. Effects of a multi-strain probiotic supplement for 12 weeks in circulating endotoxin levels and cardiometabolic profiles of medication naive T2DM patients: a randomized clinical trial. J Transl Med. 2017 Dec 11;15(1):249. doi: 10.1186/s12967-017-1354-x. PMID 29228964
- [Derived] Alokail MS, Sabico S, Al-Saleh Y, Al-Daghri NM, Alkharfy KM, Vanhoutte PM, McTernan PG. Effects of probiotics in patients with diabetes mellitus type 2: study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2013 Jul 4;14:195. doi: 10.1186/1745-6215-14-195. PMID 23822518